CLINICAL TRIAL: NCT01402284
Title: Carfilzomib, Lenalidomide, and Dexamethasone in Newly Diagnosed Multiple Myeloma: Clinical and Correlative Phase II Study
Brief Title: Carfilzomib, Lenalidomide, and Dexamethasone in New Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Celgene (Industry); Onyx Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Dickran Kazandjian, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110221; 11-C-0221
Record Dates: First submitted 2011-07-23; First posted 2011-07-26 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: Novel Drug Combinations; Protease Inhibitors; Decreased Peripheral Neuropathy; Auto Stem Cell Transplant; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib, Lenalidomide, Dexamethasone (Experimental): Patients will receive 8 cycles of induction combination therapy of carfilzomib, lenalidomide, and dexamethasone (CRd). Patients achieving stable disease or better after 8 cycles of CRd will receive lenalidomide extended dosing (phase I) for 12 cycles. After 12 cycles, patients will have the option to continue extended dosing (phase II) for one additional year
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Cycle 1: 20 mg/m(2) intravenous (IV) infusion over 30 minutes on days 1 and 2, then 36 mg/m(2) IV on days 8, 9, 15, and 16 Cycle 2-8: 36mg/ m(2) IV infusion over 30 minutes on days 1, 2, 8, 9, 15, and 16
  Other Names: Kyprolis
Drug: Lenalidomide — Cycle 1: 25 mg oral days 2-21 of 28-day cycle; Cycle 2 - 8: 25 mg oral days 1-21 of 28-day cycle; After 8 cycles of combination carfilzomib, lenalidomide, and dexamethasone (CRd), patients may continue Lenalidomide for 12 cycles; After 12 cycles of extended dosing of Lenalidomide, patients may continue Lenalidomide for one year
  Other Names: Revlimid
Drug: Dexamethasone — Cycle 1: 20 mg oral or IV on days 2, 8, 9, 15, 16, 22, and 23 Cycle 2-4: 20 mg oral or IV on days 1, 2, 8, 9, 15, 16, 22, and 23 Cycle 5-8: 10 mg oral or IV on days 1, 2, 8, 9, 15, 16, 22, and 23
  Other Names: Ozurdex
Drug: Lenalidomide — After 8 cycles of combination carfilzomib, lenalidomide, and dexamethasone (CRd), patients may continue Lenalidomide for 12 cycles
  Other Names: Revlimid
Drug: Lenalidomide — After 12 cycles of extended dosing of Lenalidomide, patients may continue Lenalidomide for one year
  Other Names: Revlimid

SUMMARY:
Background:

- Carfilzomib is an experimental anti-cancer drug that has not yet been approved for treating multiple myeloma. Lenalidomide is a drug that may stop tumor growth and help the immune system kill cancer cells. Dexamethasone is a drug that helps stop inflammation. It is sometimes used to treat (alone or with other drugs) certain types of cancer, especially multiple myeloma. This combination of drugs has not been tested in people with multiple myeloma. Researchers want to see whether it is safe and effective for this group.

Objectives:

- To test the effectiveness of combined carfilzomib, lenalidomide, and dexamethasone in treating multiple myeloma.

Eligibility:

- People at least 18 years of age who have multiple myeloma that has not been treated.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine tests, a bone marrow sample, and molecular imaging studies.
* Participants will have eight 28-day cycles of treatment. The combined study drugs will be given as tablets and injections. Those in the study will be monitored with frequent blood tests, bone marrow samples, and molecular imaging studies. In addition to current standard measures to determine clinical responses, molecular tests will be conducted to define evidence of minimal residual disease.
* After the first four cycles of therapy, those who are eligible for a stem cell transplant will have stem cells collected and stored for use if the cancer returns.
* After stem cell collection, participants will have the second four treatment cycles.

  -, If the disease has improved or is stable at the end of eight cycles, those in the study may have another 12 cycles of low-dose (maintenance) lenalidomide alone.
* Participants will have regular follow-up visits after the end of the study chemotherapy.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is an incurable plasma cell neoplasm with a median survival of 3-4 years.
* Novel agent combinations with proteasome inhibitors demonstrate improved response rates while increasing survival in MM patients.
* A common debilitating side effect of the proteasome inhibitor bortezomib is neuropathy.
* Carfilzomib is a new proteasome inhibitor with potent anti-MM effects and decreased peripheral neuropathy

Objectives:

-Evaluate toxicity, including peripheral neuropathy, of carfilzomib, lenalidomide, and dexamethasone (CRd) in untreated MM patients

Eligibility:

* Newly diagnosed patients with histologically confirmed multiple myeloma
* Age greater than or equal to 18 years
* Creatinine Clearance (CrCl) greater than or equal to 60 ml/min. CrCl will be calculated using the Cockcroft- Gault method. If the calculated CrCl based on Cockcroft-Gault method is <60 mL/min, patient will have a 24 hr urine collection to measure CrCl. The measured CrCl must also be greater than or equal to 60 ml/min.
* Without serious co-morbidity that would interfere with receipt of CRd
* Absolute neutrophil count (ANC) greater than or equal to 1.0 K/uL, hemoglobin greater than or equal to 8 g/dL, and platelet count greater than or equal to 75 K/uL
* Adequate hepatic function, with bilirubin less than 1.5 x the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3.0 x ULN

Design:

* Single arm, single stage phase II trial of combination therapy (carfilzomib, lenalidomide, and dexamethasone) for untreated multiple myeloma patients with an early stopping rule for toxicity
* Patients will receive 8 cycles of induction combination therapy of CRd
* Each cycle consists of 28-days
* After 4 cycles of therapy, transplant eligible patients will undergo stem cell collection
* Patients achieving stable disease or better after 8 cycles of CRd will receive lenalidomide extended dosing (phase I) for 12 cycles. After 12 cycles, patients will have the option to continue extended dosing (phase II) for one additional year.
* Patients will have routine blood work with serum protein electrophoresis (SPEP) and free light chains monthly
* Pre- and post-treatment bone marrow biopsies will be obtained for confirmation of diagnosis and correlative studies
* Patients will also undergo evaluation for minimal residual disease at regular interval time points, using multi-parametric flow cytometry and fludeoxyglucose 18F-positron emission tomography - computed tomography (FDG PET-CT)
* A single stage phase II design will be employed, with an early stopping rule. Unless 4 or more patients in the first 20 have Grade 3 or higher neurologic toxicity in the first 2 completed cycles, a total of 45 evaluable patients will be enrolled in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Newly diagnosed patients with histologically confirmed multiple myeloma (MM) based on the following criteria:

  1. Clonal plasma cells in the bone marrow
  2. Measurable disease within the past 4 weeks defined by any one of the following:

     1. Serum monoclonal protein greater than or equal to 1.0 g/dL
     2. Urine monoclonal protein greater than 200 mg/24 hour
     3. Serum immunoglobulin free light chain greater than 10 mg/dL AND abnormal kappa/lambda ratio
  3. Evidence of underlying end organ damage attributed to underlying plasma cell proliferative disorder meeting at least one of the following:

     1. Hypercalcemia: serum calcium greater than or equal to 2.65 mmol/L
     2. Renal Insufficiency: serum creatinine greater than 2.0 mg/dL
     3. Anemia: hemoglobin value less than10 g/dL or 2 g/dL less than normal reference
     4. Bone disease: lytic lesions, severe osteopenia or pathological fractures
* Creatinine Clearance (CrCl) greater than or equal to 60 ml/min. CrCl will be calculated by Cockcroft-Gault method. CrCl (calculated) = (140 Age) x Mass (in kilograms) x [0.85 if Female] 72 times Serum Creatinine (in mg/dL). If calculated CrCl based on Cockcroft-Gault method is <60 mL/min, patient will have a 24 hr urine collection to measure CrCl. The measured CrCl must be also greater than or equal to 60 ml/min.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of carfilzomib in combination with lenalidomide in patients less than18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) greater than or equal to 1.0 K/uL, hemoglobin greater than or equal to 8 g/dL (transfusions are permissible), and platelet count greater than or equal to 75 K/uL
* Adequate hepatic function, with bilirubin less than 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3.0 times ULN.
* All study participants must be able to tolerate one of the following thromboprophylactic strategies: aspirin, low molecular weight heparin or warfarin (coumadin).
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist .
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 10-14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. Females of child bearing potential (FCBP) must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Subjects must be able to give informed consent

EXCLUSION CRITERIA:

* Prior or concurrent systemic treatment for MM.

  * Treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with corticosteroids is permitted.
  * Bisphosphonates are permitted.
  * Treatment with corticosteroids for indications other than MM is permitted.
  * Radiotherapy is permitted.
  * Treatment for smoldering myeloma is permitted.
* Plasma cell leukemia
* Pregnant or lactating females. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with carfilzomib in combination with lenalidomide, breastfeeding should be discontinued if the mother is treated with carfilzomib and lenalidomide. These potential risks may also apply to other agents used in this study.
* Uncontrolled hypertension or diabetes
* Active hepatitis B or C infection
* Has significant cardiovascular disease with New York Heart Association (NYHA) Class III or IV symptoms, or hypertrophic cardiomyopathy, or restrictive cardiomyopathy, or myocardial infarction within 3 months prior to enrollment, or unstable angina, or unstable arrhythmia as determined by history and physical examination. Echocardiogram will be performed if clinically warranted.
* Has refractory gastrointestinal (GI) disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption
* Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance with study requirements
* Significant neuropathy greater than or equal to Grade 3 at baseline
* Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy
* Major surgery within 1 month prior to enrollment
* Recruitment Strategies:

  * Patients that progress from the smoldering multiple myeloma (SMM) and monoclonal gammopathy of undetermined significance (MGUS) Natural History Study (NCI Protocol: 10-C-0096) will be potential candidates.
  * Other participant sources will be from outside physician referrals.
  * Our ongoing natural history study and outside physician referral network has a high representation of minorities.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-07-21 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dickran Kazandjian, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Myeloma Working Group. Criteria for the classification of monoclonal gammopathies, multiple myeloma and related disorders: a report of the International Myeloma Working Group. Br J Haematol. 2003 Jun;121(5):749-57. PMID 12780789
- [Background] Kristinsson SY, Landgren O, Dickman PW, Derolf AR, Bjorkholm M. Patterns of survival in multiple myeloma: a population-based study of patients diagnosed in Sweden from 1973 to 2003. J Clin Oncol. 2007 May 20;25(15):1993-9. doi: 10.1200/JCO.2006.09.0100. Epub 2007 Apr 9. PMID 17420512
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Derived] Landgren O, Kazandjian D, Roussel M, Jasielec J, Dytfeld D, Anderson A, Kervin TA, Iskander K, McFadden I, Jakubowiak AJ. Efficacy and safety of carfilzomib-lenalidomide-dexamethasone in newly diagnosed multiple myeloma: pooled analysis of four single-arm studies. Leuk Lymphoma. 2022 Oct;63(10):2413-2421. doi: 10.1080/10428194.2022.2068001. Epub 2022 May 12. PMID 35549810
- [Derived] Huang PA, Beedie SL, Chau CH, Venzon DJ, Gere S, Kazandjian D, Korde N, Mailankody S, Landgren O, Figg WD. Cereblon gene variants and clinical outcome in multiple myeloma patients treated with lenalidomide. Sci Rep. 2019 Oct 16;9(1):14884. doi: 10.1038/s41598-019-51446-9. PMID 31619706
- [Derived] Acosta-Alvear D, Cho MY, Wild T, Buchholz TJ, Lerner AG, Simakova O, Hahn J, Korde N, Landgren O, Maric I, Choudhary C, Walter P, Weissman JS, Kampmann M. Paradoxical resistance of multiple myeloma to proteasome inhibitors by decreased levels of 19S proteasomal subunits. Elife. 2015 Sep 1;4:e08153. doi: 10.7554/eLife.08153. PMID 26327694
- [Derived] Korde N, Roschewski M, Zingone A, Kwok M, Manasanch EE, Bhutani M, Tageja N, Kazandjian D, Mailankody S, Wu P, Morrison C, Costello R, Zhang Y, Burton D, Mulquin M, Zuchlinski D, Lamping L, Carpenter A, Wall Y, Carter G, Cunningham SC, Gounden V, Sissung TM, Peer C, Maric I, Calvo KR, Braylan R, Yuan C, Stetler-Stevenson M, Arthur DC, Kong KA, Weng L, Faham M, Lindenberg L, Kurdziel K, Choyke P, Steinberg SM, Figg W, Landgren O. Treatment With Carfilzomib-Lenalidomide-Dexamethasone With Lenalidomide Extension in Patients With Smoldering or Newly Diagnosed Multiple Myeloma. JAMA Oncol. 2015 Sep;1(6):746-54. doi: 10.1001/jamaoncol.2015.2010. PMID 26181891
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0221.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Carfilzomib, Lenalidomide, and Dexamethasone Therapy: Patients will receive 8 cycles of induction combination therapy of carfilzomib, lenalidomide, and dexamethasone (CRd). Patients achieving stable disease or better after 8 cycles of CRd will receive lenalidomide extended dosing (phase I) for 12 cycles. After 12 cycles, patients will have the option to continue extended dosing (phase II) for one additional year Carfilzomib: Cycle 1: 20 mg/m(2) intravenous (IV) infusion over 30 minutes on days 1 and 2, then 36 mg/m(2) IV on days 8, 9, 15, and 16 Cycle 2-8: 36mg/ m(2) IV infusion over 30 minutes on days 1, 2, 8, 9, 15, and 16 Lenalidomide: Cycle 1: 25 mg oral days 2-21 of 28-day cycle; Cycle 2 - 8: 25 mg oral days 1-21 of 28-day cycle; After 8 cycles of combination carfilzomib, lenalidomide, and dexamethasone (CRd), patients may continue Lenalidomide for 12 cycles; After 12 cycles of extended dosing of Lenalidomide, patients may continue Lenalidomide for one year Dexamethasone: Cycle 1: 20 mg oral or IV on days 2, 8, 9, 15, 16, 22,
Period: Overall Study
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone Therapy
Started | 45
Completed | 31
Not Completed | 14
Not completed — Withdrawal consent | 2
Not completed — Follows up at Memorial Sloan Kettering | 1
Not completed — Physician Decision | 1
Not completed — Disease progression on study | 10

BASELINE CHARACTERISTICS:
Groups:
- Carfilzomib, Lenalidomide, and Dexamethasone: Patients will receive 8 cycles of induction combination therapy of carfilzomib, lenalidomide, and dexamethasone (CRd). Patients achieving stable disease or better after 8 cycles of CRd will receive lenalidomide extended dosing (phase I) for 12 cycles. After 12 cycles, patients will have the option to continue extended dosing (phase II) for one additional year Carfilzomib: Cycle 1: 20 mg/m(2) intravenous (IV) infusion over 30 minutes on days 1 and 2, then 36 mg/m(2) IV on days 8, 9, 15, and 16 Cycle 2-8: 36mg/ m(2) IV infusion over 30 minutes on days 1, 2, 8, 9, 15, and 16 Lenalidomide: Cycle 1: 25 mg oral days 2-21 of 28-day cycle; Cycle 2 - 8: 25 mg oral days 1-21 of 28-day cycle; After 8 cycles of combination carfilzomib, lenalidomide, and dexamethasone (CRd), patients may continue Lenalidomide for 12 cycles; After 12 cycles of extended dosing of Lenalidomide, patients may continue Lenalidomide for one year Dexamethasone: Cycle 1: 20 mg oral or IV on days 2, 8, 9, 15, 16, 22,
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45
Isotypes [Number; unit: percentage of participants] — Measure Description: IgA Kappa, IgG Kappa, IgG Lambda, Free Kappa and Free lambda were measured in the urine to determine changes in renal function. Measurable is defined as any of the following: Serum monoclonal protein greater than or equal to 1.0 g/dL, urine monoclonal protein greater than 200 mg/24 hour, and serum immunoglobulin free light chain greater than 10mg/dL AND abnormal kappa/lambda ratio.
  percentage of participants
    IgG kappa | 51
    IgG lambda | 16
    IgA kappa | 9
    IgA lambda | 9
    Free kappa | 9
    Free lambda | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 4 years and 9 months and 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
Participants | 45

2. Secondary Outcome: Overall Response Rate
Description: Response is assessed by the International Myeloma Working Group Criteria. Patients who attained a partial response or better (BoR) response by the end of induction. Partial response is ≥50% reduction of serum M-protein and reduction in 24h urinary M-protein.
Time Frame: 48.3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
percentage of participants | 97.8 [88.2 to 99.9]

3. Secondary Outcome: Progression Free Survival (PFS) at 48 Months
Description: PFS is defined as time of start of treatment to time of progression or death, whichever occurs first. Response is assessed by the International Myeloma Working Group Criteria. Progressive disease requires any one or more of the following: increase of ≥25% from lowest response value in the following on 2 consecutive measurements: serum M-component and/or (the absolute increase must be ≥0.5g/dl). Urine M-component and/or (the absolute increase must be ≥200mg/24h. Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels. The absolute increase must be >10mg/dl. Bone marrow plasma cell percentage: the absolute % must be ≥10%. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: 48 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
percentage of participants | 79.2 [63.8 to 88.6]

4. Secondary Outcome: Percentage of Responders With Duration of Response (DOR) at 48 Months
Description: Response is assessed by the International Myeloma Working Group Criteria. DOR is measured from the time measurement criteria are met for a partial response or better until first date that recurrent or progressive disease is objectively documented. Partial response is ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200mg per 24h. Progressive disease requires any one or more of the following: increase of ≥25% from lowest response value in the following on 2 consecutive measurements: serum M-component and/or (the absolute increase must be ≥0.5g/dl). Urine M-component and/or (the absolute increase must be ≥200mg/24h. Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels. The absolute increase must be >10mg/dl. Bone marrow plasma cell percentage: the absolute % must be ≥10%.
Time Frame: 48 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
percentage of participants | 81.1 [65.7 to 90.1]

5. Secondary Outcome: Overall Survival (OS) Rate
Description: OS is defined as the time of start of treatment to death from any cause.
Time Frame: up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
percentage of participants | 89.5 [63.6 to 97.3]

6. Secondary Outcome: Cluster of Differentiation 138 (CD138) + Plasma Cells Gene Expression Profiling on Pre and Post Carfilzomib Exposure Bone Marrow Samples
Description: Cluster of differentiation 138+ (CD138)+ plasma cells purified from bone marrow aspirates to identify potential markers of early progression. Changes in selected genes were confirmed by quantitative polymerase chain reaction (PCR) if suggested to be related to risk of progression to multiple myeloma.
Time Frame: Cycle 1 Day 1, an average of 28 days ± 2 days
Population: Data were not collected due to lack of financial resources.
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of Minimal Residual Disease (MRD) by Flow Cytometry
Description: Response is assessed by the International Myeloma Working Group Criteria. Complete response is negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow. MRD is defined by M-spike, plasma cell burden, and abnormal free light chains. Immunophenotyping is performed by multi-parametric flow cytometry.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
percentage of participants | 44.4 [29.6 to 60.0]

8. Secondary Outcome: Complete Response (CR) and Minimal Residual Disease Neg (MRDneg) CR Rates at Treatment Intervals With Carfilzomib, Lenalidomide & Dexamethasone (CRd) in New Multiple Myeloma Patients After 8 Cycles of Induction, 1 Year Maintenance, and 2 Years Maintenance
Description: Response is assessed by the International Myeloma Working Group Criteria. MRD is defined by M-spike, plasma cell burden, and abnormal free light chains (FLC). Complete response is negative immunofixation on serum, and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow. Stringent complete response (sCR) is normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence. Near complete response (nCR) is the absence of myeloma protein on electrophoresis, independent of immunofixation status. Very good partial response (VGPR) is serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24h. Overall response rate (ORR) is patients who attained a partial response (PR) (≥50% reduction of serum M-protein and reduction in 24h urinary M-protein) or better (BoR) response.
Time Frame: up to 2 years
Population: *Six patients withdrew from the study, four due to non-compliance and two to continue treatment at another institution. 'One patient refused to have a bone marrow biopsy procedure and one patient withdrew due to non-compliance. CR (n=0) after 8 cycles.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
Number analyzed (Participants) | 45
percentage of participants
  sCR/CR after 8 cycles: number analyzed (Participants) | 21
  sCR/CR after 8 cycles | 46.7 [31.7 to 62.1]
  MRDnegCR after 8 cycles: number analyzed (Participants) | 20
  MRDnegCR after 8 cycles | 44.4 [29.6 to 60.0]
  nCR after 8 cycles: number analyzed (Participants) | 9
  nCR after 8 cycles | 20 [9.6 to 34.6]
  ≥VGPR after 8 cycles: number analyzed (Participants) | 40
  ≥VGPR after 8 cycles | 89 [75.6 to 96.3]
  ORR after 8 cycles: number analyzed (Participants) | 44
  ORR after 8 cycles | 97.8 [88.2 to 99.9]
  sCR after 8 cycles: number analyzed (Participants) | 21
  sCR after 8 cycles | 46.7 [31.7 to 62.1]
  sCR/CR after 1 year: number analyzed (Participants) | 28
  sCR/CR after 1 year | 62.2 [46.5 to 76.2]
  sCR after 1 year: number analyzed (Participants) | 27
  sCR after 1 year | 60.0 [44.3 to 74.3]
  CR after 1 year: number analyzed (Participants) | 1
  CR after 1 year | 2.2 [0 to 11.8]
  MRDnegCR after 1 year': number analyzed (Participants) | 23
  MRDnegCR after 1 year' | 53.5 [37.7 to 68.8]
  nCR after 1 year: number analyzed (Participants) | 5
  nCR after 1 year | 11.1 [3.7 to 24.1]
  ≥VGPR after 1 year: number analyzed (Participants) | 40
  ≥VGPR after 1 year | 89 [75.6 to 96.3]
  ORR after 1 year: number analyzed (Participants) | 44
  ORR after 1 year | 97.8 [88.2 to 99.9]
  sCR/CR after 2 years: number analyzed (Participants) | 29
  sCR/CR after 2 years | 64.4 [48.8 to 78.1]
  sCR after 2 years: number analyzed (Participants) | 28
  sCR after 2 years | 62.2 [46.5 to 76.2]
  CR after 2 years: number analyzed (Participants) | 1
  CR after 2 years | 2.2 [0 to 11.8]
  MRDnegCR after 2 years*: number analyzed (Participants) | 18
  MRDnegCR after 2 years* | 46.2 [30.1 to 62.8]
  nCR after 2 years: number analyzed (Participants) | 5
  nCR after 2 years | 11.1 [3.7 to 24.1]
  ≥VGPR after 2 years: number analyzed (Participants) | 41
  ≥VGPR after 2 years | 91.1 [78.8 to 97.5]
  ORR after 2 years: number analyzed (Participants) | 44
  ORR after 2 years | 97.8 [88.2 to 99.9]

ADVERSE EVENTS:
Time Frame: 4 years and 9 months and 2 days
Arm/Group | Carfilzomib, Lenalidomide, and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 3/45
Serious Adverse Events (participants affected / at risk) | 19/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib, Lenalidomide, and Dexamethasone (N=45)
Adrenal insufficiency (Endocrine disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (8)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (3)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Edema limbs (General disorders) | 2 (2)
Enterocolitis infectious (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (3)
Fever (General disorders) | 3 (3)
General disorders and administration site conditions - Other, night sweats/tremors (General disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 6 (6)
White blood cell decreased (Investigations) | 1 (1)
Death (General disorders) | 2 (45)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib, Lenalidomide, and Dexamethasone (N=45)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 7 (9)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 36 (166)
Alkaline phosphatase increased (Investigations) | 29 (67)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 34 (148)
Anorexia (Metabolism and nutrition disorders) | 5 (7)
Anxiety (Psychiatric disorders) | 3 (5)
Appendicitis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 25 (71)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 23 (72)
Blurred vision (Eye disorders) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
CPK increased (Investigations) | 10 (19)
Cardiac disorders - Other, cardiac NOS (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 11 (14)
Chills (General disorders) | 5 (6)
Cognitive disturbance (Nervous system disorders) | 4 (4)
Concentration impairment (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Creatinine increased (Investigations) | 18 (51)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 30 (51)
Dizziness (Nervous system disorders) | 4 (4)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (37)
Edema face (General disorders) | 4 (5)
Edema limbs (General disorders) | 17 (30)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
Enterocolitis infectious (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 8 (9) — Diminished visual; diplopia; visual changes; conjunctival bleeding L eye; increased intraocular pressure; scleral redness
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 28 (43)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 12 (18)
Flu like symptoms (General disorders) | 5 (5)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (8)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Gastrointeritis (General disorders) | 1 (1)
Generalized muscle weakness (General disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Glaucoma (Eye disorders) | 2 (2)
Headache (Nervous system disorders) | 15 (21)
Heart failure (Cardiac disorders) | 2 (2)
Hematoma (Vascular disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hot flashes (Vascular disorders) | 6 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 10 (18)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (12)
Hypermagnesemia (Metabolism and nutrition disorders) | 23 (35)
Hypernatremia (Metabolism and nutrition disorders) | 26 (52)
Hypertension (Vascular disorders) | 5 (16)
Hyperuricemia (Metabolism and nutrition disorders) | 12 (25)
Hypoalbuminemia (Metabolism and nutrition disorders) | 42 (136)
Hypocalcemia (Metabolism and nutrition disorders) | 20 (36)
Hypokalemia (Metabolism and nutrition disorders) | 10 (19)
Hypomagnesemia (Metabolism and nutrition disorders) | 17 (40)
Hyponatremia (Metabolism and nutrition disorders) | 16 (33)
Hypophosphatemia (Metabolism and nutrition disorders) | 29 (79)
Hypotension (Vascular disorders) | 2 (3)
Hypothyroidism (Endocrine disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) — Cellulitis' cellulitis L. ankle; flu; zoster
Infusion related reaction (General disorders) | 3 (5)
Injection site reaction (General disorders) | 32 (51)
Insomnia (Psychiatric disorders) | 26 (30)
Irritability (General disorders) | 4 (4)
Laryngitis (Infections and infestations) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (2)
Lipase increased (Investigations) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (4)
Lymphocyte count decreased (Investigations) | 45 (438)
Lymphocyte count increased (Investigations) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 6 (9) — Achilles; bursitis; cramps/hands; cramps/legs; leg cramps; R rotator cuff tear; trigger finger R hand; umbilical hernia repair
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (19)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — BCC; papillary urothelial neoplasm
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 35 (207)
Nocturia (Renal and urinary disorders) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Pain (General disorders) | 19 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (17)
Palpitations (Cardiac disorders) | 3 (3)
Papilledema (Eye disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 22 (33)
Personality change (Psychiatric disorders) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2)
Platelet count decreased (Investigations) | 42 (214)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8)
Psychiatric disorders - Other, Emotional lability (Psychiatric disorders) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 (68)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Rhinorrhea; Rt. Pleural density (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis infective (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Sinusitis (Infections and infestations) | 5 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (5) — L. foot ruddy and taut; scalp sensitivity; skin lesion RLE; squamous cell skin cancer L thigh; sunburn
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (6)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Tremor (Nervous system disorders) | 9 (11)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 30 (47)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular disorders - Other, Raynaud's disorder (Vascular disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 38 (284)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT01402284/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT01402284/ICF_003.pdf